CLINICAL TRIAL: NCT00236301
Title: Pro-Inflammatory Effects of Two Different Doses of 17 Beta Estradiol in Menopausal Women
Brief Title: Dose Effects of Hormone Therapy (Two Doses of Estradiol Associated to Progesterone) on Inflammatory Markers
Acronym: THS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: terminated
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: French Health Products Safety Agency (Other Government); FRM (Unknown); Solvay Pharmaceuticals (Industry)
Responsible Party: Yannick Vacher, Department Clinical Research of Developement
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P021204
Record Dates: First submitted 2005-10-11; First posted 2005-10-12 (Estimated); Last update posted 2008-01-17 (Estimated); Status verified 2005-10

CONDITIONS: Healthy Symptomatic Menopausal Women
Keywords: Hormone; Menopause; Inflammation; Dose effects; Apoptosis
MeSH Terms: conditions — Inflammation | interventions — Pharmaceutical Preparations; Estradiol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Active Comparator): 17 Beta-estradiol (2mg/day)and (1mg/day)
  Interventions: Drug: 17 Beta-estradiol (2mg/day)and (1mg/day)
- 2 (Active Comparator): CLIMASTON
  Interventions: Drug: CLIMASTON (drug)
- 3 (Placebo Comparator): placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: CLIMASTON (drug) — CLIMASTON(drug)
  Arms: 2
Drug: 17 Beta-estradiol (2mg/day)and (1mg/day) — 17 Beta-estradiol (2mg/day)and (1mg/day)
  Arms: 1
Drug: placebo — placebo
  Arms: 3

SUMMARY:
Primary purpose : Effects of two doses of hormone therapy on hsCRP. The effects of hormone replacement therapy on inflammatory markers are dose-dependent.

DETAILED DESCRIPTION:
Pro-inflammatory study of the effects in short term of two difference doses of 17beta-estradiol at the menopause woman

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic menopausal women : >=50 years and amenorrhea >=1 year or <50 years and amenorrhea >=1 year and plasmatic FSH >= 30 UI/l
* Normal mammography in the last 2 years before inclusion
* Normal cervical smear in the last 2 years before inclusion
* Written consent for participation in the study

Exclusion Criteria:

* Unconfirmed Menopause with amenorrhoea of less than year
* Oestrogen-progesterone Treatment anterior in 3 months previous the inclusion
* Recently a viral Infection or bacteriologic(at least of 2 weeks)
* Dental Infection
* Inflammatory Pathology chronicles
* Antecedent of pathology cancerous with or no a sly hemopathy
* Addiction to smoking of more than 20 cigarettes a day or an alcoholic consumption furthermore of 4 glasses a day
* Taken concomitant of one of the treatments forbidden:statine, vitamin B6 or B12, folates, antiinflammatory, anti aggregant Plaquettes, DHEA, phytoestrogens
* Refusal to sign the assent informed
* Not membership in a regime about social security

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2004-03; Primary Completion 2006-06 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Hs-C-reactive protein | 2 months

SECONDARY OUTCOMES:
Interleukin (IL-6, IL-18, IL-10), TNF-alpha, apoptotic microparticles, homocysteine, total cholesterol/HDL cholesterol, Lp(a), interleukin 6, ICAM soluble, | 2 months
Eslectin, prothrombin F1+2, factor VIII, resistance to activated protein C (RPCA or ACV test),IL 18, IL10, IL8 | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Tabassome Simon, M.D., Ph.D., Principal Investigator — Service de Pharmacologie (Pr Jaillon) CHU Saint-Antoine 27, rue de Chaligny, 75012 Paris
Locations (1):
- CIC, Saint Antoine Hospital, Paris, France

REFERENCES:
- [Background] Colditz GA, Willett WC, Stampfer MJ, Rosner B, Speizer FE, Hennekens CH. Menopause and the risk of coronary heart disease in women. N Engl J Med. 1987 Apr 30;316(18):1105-10. doi: 10.1056/NEJM198704303161801. PMID 3574358
- [Background] Hodis HN, Mack WJ, Lobo RA, Shoupe D, Sevanian A, Mahrer PR, Selzer RH, Liu Cr CR, Liu Ch CH, Azen SP; Estrogen in the Prevention of Atherosclerosis Trial Research Group. Estrogen in the prevention of atherosclerosis. A randomized, double-blind, placebo-controlled trial. Ann Intern Med. 2001 Dec 4;135(11):939-53. doi: 10.7326/0003-4819-135-11-200112040-00005. PMID 11730394
- [Background] Rossouw JE, Anderson GL, Prentice RL, LaCroix AZ, Kooperberg C, Stefanick ML, Jackson RD, Beresford SA, Howard BV, Johnson KC, Kotchen JM, Ockene J; Writing Group for the Women's Health Initiative Investigators. Risks and benefits of estrogen plus progestin in healthy postmenopausal women: principal results From the Women's Health Initiative randomized controlled trial. JAMA. 2002 Jul 17;288(3):321-33. doi: 10.1001/jama.288.3.321. PMID 12117397
- [Background] Mendelsohn ME, Karas RH. The protective effects of estrogen on the cardiovascular system. N Engl J Med. 1999 Jun 10;340(23):1801-11. doi: 10.1056/NEJM199906103402306. No abstract available. PMID 10362825
- [Background] Scarabin PY, Alhenc-Gelas M, Plu-Bureau G, Taisne P, Agher R, Aiach M. Effects of oral and transdermal estrogen/progesterone regimens on blood coagulation and fibrinolysis in postmenopausal women. A randomized controlled trial. Arterioscler Thromb Vasc Biol. 1997 Nov;17(11):3071-8. doi: 10.1161/01.atv.17.11.3071. PMID 9409295
- [Background] Teede HJ, McGrath BP, Smolich JJ, Malan E, Kotsopoulos D, Liang YL, Peverill RE. Postmenopausal hormone replacement therapy increases coagulation activity and fibrinolysis. Arterioscler Thromb Vasc Biol. 2000 May;20(5):1404-9. doi: 10.1161/01.atv.20.5.1404. PMID 10807761
- [Background] Conard J, Basdevant A, Thomas JL, Ochsenbein E, Denis C, Guyene TT, Degrelle H. Cardiovascular risk factors and combined estrogen-progestin replacement therapy: a placebo-controlled study with nomegestrol acetate and estradiol. Fertil Steril. 1995 Nov;64(5):957-62. doi: 10.1016/s0015-0282(16)57909-6. PMID 7589641
- [Background] Ridker PM, Hennekens CH, Buring JE, Rifai N. C-reactive protein and other markers of inflammation in the prediction of cardiovascular disease in women. N Engl J Med. 2000 Mar 23;342(12):836-43. doi: 10.1056/NEJM200003233421202. PMID 10733371
- [Background] Mallat Z, Heymes C, Ohan J, Faggin E, Leseche G, Tedgui A. Expression of interleukin-10 in advanced human atherosclerotic plaques: relation to inducible nitric oxide synthase expression and cell death. Arterioscler Thromb Vasc Biol. 1999 Mar;19(3):611-6. doi: 10.1161/01.atv.19.3.611. PMID 10073964
- [Background] Mallat Z, Hugel B, Ohan J, Leseche G, Freyssinet JM, Tedgui A. Shed membrane microparticles with procoagulant potential in human atherosclerotic plaques: a role for apoptosis in plaque thrombogenicity. Circulation. 1999 Jan 26;99(3):348-53. doi: 10.1161/01.cir.99.3.348. PMID 9918520
- [Background] Mallat Z, Benamer H, Hugel B, Benessiano J, Steg PG, Freyssinet JM, Tedgui A. Elevated levels of shed membrane microparticles with procoagulant potential in the peripheral circulating blood of patients with acute coronary syndromes. Circulation. 2000 Feb 29;101(8):841-3. doi: 10.1161/01.cir.101.8.841. PMID 10694520
- [Background] Ridker PM, Hennekens CH, Rifai N, Buring JE, Manson JE. Hormone replacement therapy and increased plasma concentration of C-reactive protein. Circulation. 1999 Aug 17;100(7):713-6. doi: 10.1161/01.cir.100.7.713. PMID 10449692
- [Background] Cushman M, Legault C, Barrett-Connor E, Stefanick ML, Kessler C, Judd HL, Sakkinen PA, Tracy RP. Effect of postmenopausal hormones on inflammation-sensitive proteins: the Postmenopausal Estrogen/Progestin Interventions (PEPI) Study. Circulation. 1999 Aug 17;100(7):717-22. doi: 10.1161/01.cir.100.7.717. PMID 10449693
- [Background] Scarabin PY, Alhenc-Gelas M, Oger E, Plu-Bureau G. Hormone replacement therapy and circulating ICAM-1 in postmenopausal women--a randomised controlled trial. Thromb Haemost. 1999 May;81(5):673-5. PMID 10365734
- [Background] van Baal WM, Smolders RG, van der Mooren MJ, Teerlink T, Kenemans P. Hormone replacement therapy and plasma homocysteine levels. Obstet Gynecol. 1999 Oct;94(4):485-91. doi: 10.1016/s0029-7844(99)00412-3. PMID 10511346